CLINICAL TRIAL: NCT02605980
Title: The Acute Effects of Sitting Time on Physiological and Psychological Function in Older Adults
Brief Title: Acute Effects of Sitting Time in Older Adults
Acronym: ACUSIT
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: The Dunhill Medical Trust (Other); Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Other Study IDs: 177149
Record Dates: First submitted 2015-10-16; First posted 2015-11-17 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2016-03

CONDITIONS: Ageing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and serum from living donors
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Male: Community-dwelling healthy older adults over the age of 70 years. Must be ambulatory, with or without walking aids
  Interventions: Behavioral: Sedentary time
- Female: Community-dwelling healthy older adults over the age of 70 years. Must be ambulatory, with or without walking aids
  Interventions: Behavioral: Sedentary time

INTERVENTIONS:
Behavioral: Sedentary time

SUMMARY:
United Kingdom (UK) physical activity guidelines for older people state that "All older adults should minimise the amount of time spent being sedentary (sitting) for extended periods" and "there is sufficient evidence to support a recommendation to reduce sedentary behaviour in older adults, but it is not currently possible to suggest a specific time limit." The aim of this study is to identify key physiological and psychological outcomes influenced by acute periods of inactivity and what older people feel after these acute periods of inactivity. The investigators' main objective is to determine, through direct measurement and self report, the acute functional and cognitive effects of differing periods of sitting time. A secondary objective is to inform older people, professionals and organisations working with older people and policy makers on what duration of sedentary behaviour will lead to adverse outcomes in older people. The investigators will recruit ambulatory men and women aged 70 y and over who will be studied on three separate occasions, approximately one week apart to complete sedentary bouts of 1 h, 2 h and 4 h in a randomised crossover design. The investigators will explore the relationship between sitting time and changes in lower limb explosive power(primary outcome) measured before and after each bout. Secondary outcomes will include timed chair rise; Timed Up and Go; blood pressure; perception of musculoskeletal comfort/pain, vitality; mood and cognitive function. The investigators will also measure the stress hormone cortisol in samples of saliva taken at the start of the sitting session, 1 h, 2h and 4 h later. Characterising the acute effects of sitting time in older adults will enable the design of interventions to reduce sedentary time as well as inform professionals and policy makers on what duration of sedentary behaviour will lead to adverse outcomes.

DETAILED DESCRIPTION:
Until relatively recently, sedentary behaviour was considered as the 'lower end' of the physical activity spectrum. However there is accumulating evidence from both epidemiological and observational studies which shows that sedentary behaviour per se rather than just low physical activity is also a major modifiable risk factor for chronic disease and predicts cardiovascular and all-cause mortality, independent of the amount of physical activity: A followup of the Australian Diabetic (AusDiab) cohort study showed a 46% increased risk of all-cause and an 80% increased risk of cardiovascular disease mortality in those watching four or more hours of television (TV) per day, compared with those watching TV for <2 h per day. In the Canadian Fitness Survey, a dose response relationship was shown between sitting time and cardiovascular disease and all-cause mortality. Significantly poorer long term mortality outcomes were found in those reporting spending most of the day sitting compared with those reporting less time sitting and this was consistent across all levels of self reported sitting time. Crucially, sitting time mortality relationships were apparent even among those who were physically active at other time points in their day. Although there is evidence supporting the longer term detrimental health effects of prolonged bouts of sedentary behaviour (sitting) across the age range, limited information exists with respect to the acute (or 'last bout') effects of sedentariness on the physiological and psychological health of older people.

Interestingly the current UK physical activity guidelines state that "while there is sufficient evidence to support a recommendation to reduce sedentary behaviour in older adults, it is not currently possible to suggest a specific time limit". There is the need to be able to characterise sitting time in older adults in terms of acute functional and cognitive effects, as well as identify the main effects that older people perceive as being important after periods of sitting. Thus there is a possibility of generating specific advice to older people, but this requires the elucidation of dose response relationships between sitting and health outcomes to be defined during carefully controlled studies. Although these studies have yet to be conducted, it is possible to select 'key' outcome measures based upon established evidence derived from epidemiological and smaller scale observational studies (viz recent studies reporting a significant negative association between sedentariness and physical and psychological impairment in older adults) as well as from other 'models' of physical inactivity such as bed rest and limb unloading. One such outcome is skeletal muscle power output. The ability to quickly produce sufficient muscle power is of paramount importance for controlling body movements during mobility related activities in older people, such as standing up from a chair or stair climbing. Muscle power output is therefore a functionally relevant outcome of the utmost importance to the maintenance of physical independence. In addition, older people are less able to maintain core temperature, partly due to a reduced muscle mass yet it is known that reducing muscle temperature by only 1˚C can result in a decline of power output of up to 26%. Work by the current study group has recently shown a reduction in muscle power (45%), sit to stand performance velocity (9%), gait speed and maximum quadriceps strength after only 45 minutes sitting in a cool environment (15 degrees Celsius). It is not known if sitting (and consequent muscle inactivity) in normal temperature environments leads to reduced power in older people. However, older people talk of more difficulty getting out of a chair when they have been sitting for long periods, so muscle power may be implicated. In older people with joint pain, the benefits of keeping moving and not just sitting are clear.

Although work on the effect of cold environments on cognition (dual task cost in walking speed and executive function using the trail making test) did not show any significant changes after 45 minutes exposure to 15 degrees Celsius in older people, little is known about effects on mood, well being or other cognitive and psychological outcomes of sitting. Associations between sitting and tiredness and depression have been shown in a longitudinal study of a middle aged Australian cohort in those who spent a total of >9 h/day sitting compared with those who spent <6 h/day sitting. However little is known about the effects of acute bouts of sitting. Although there is a body of evidence on the acute effects of physical activity, no published data reporting acute effects of sitting, or on dose response effects on psychological outcomes was found.

Thus, the current understanding of the acute effects of sitting time is severely limited. The proposed study will inform the development, implementation and evaluation of future interventions to reduce sedentary behaviour in older people by identifying key elements of the immediate (acute) benefits of breaking up long periods of sitting, aiding engagement with older adults about immediate individual level benefits of reduced sitting and identifying outcome measures sensitive to changes in sitting time. Alongside views of older people, it will provide practical messages that can ensure more effective take up of an intervention among older people and effective advice for the professionals that work with older people. For example, for professionals working in residential home settings or on hospital wards/ intermediate or transition care settings (post acute illness or surgery), the results of this research will give valuable information on desirable time periods for encouraging mobilisation.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or over
* Ambulatory with or without a walking aid.

Exclusion Criteria:

* History of myocardial infarction within previous 2 years
* Cardiac illness: moderate/ severe aortic stenosis, acute pericarditis, acute myocarditis, aneurysm, severe angina, clinically significant valvular disease, uncontrolled dysrhythmia, claudication within the previous 10 years
* Thrombophlebitis or pulmonary embolus within the previous 2 years
* History of cerebrovascular disease (CVA or TIA) within the previous 2 years
* Acute febrile illness within the previous 3 months
* Severe airflow obstruction
* Uncontrolled metabolic disease (e.g., thyroid disease or cancer)
* Significant emotional distress, psychotic illness or depression within the previous 2 years
* Lower limb fracture sustained within the previous 2 years; upper limb fracture within the previous 6 months; non arthroscopic lower limb joint surgery within the previous 2 years
* Any reason for loss of mobility for greater than 1 week in the previous 2 months or greater than 2 weeks in the previous 6 months
* Poorly controlled atrial fibrillation
* Poor (chronic) pain control
* Resting systolic pressure >200 mmHg or resting diastolic pressure >100 mmHg
* Moderate/ severe cognitive impairment (MMSE <23)
* Impaired tissue viability (defined by a Waterlow risk assessment score >15).

Based on Greig C.A. et al. Age Ageing 1994, 23: 185-9

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling healthy older adults aged 70 years or over. Must be ambulatory with or without a walking aid.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in lower limb extensor power (Nottingham Power Rig) | This will be assessed seven times within a period of six weeks throughout the study. First will be at the start of study (first visit).Two more tests will be conducted each time on the second,third and final visits which will be one week apart.
  The design of the device includes an adjustable seat and a footplate connected through a chain and lever to a flywheel. There is an attached seat which is adjustable to the appropriate position for each participant, ensuring that when the footplate is fully depressed, the participant's leg will be in the extended position. The participant will sit upright in the seat with arms crossed across the chest and non- dominant leg resting with the foot flat on the floor or frame of the rig. The participants will be required to apply maximal force to the footplate, by extending their dominant leg with maximal effort. When force is applied to the footplate, the flywheel accelerates, initiating the data collection. The final velocity of the flywheel will be used to calculate power (W.kg-1), which will then be displayed on a computer interface.

SECONDARY OUTCOMES:
Change in Timed chair rise (functional ability) | This will be assessed seven times across three sessions (one week apart) over a period of six weeks throughout the study i.e.at the start of study, and two more tests each time on the second,third and final visits.
  This is a measure of the time taken for each participant to rise from sitting on a chair to upright standing.
Change in Timed Up and Go (marker of falls risk) | This measure will be assessed seven times across three sessions (one week apart) over a period of six weeks throughout the study period.
  This test involves instructing the participants to stand from a seated position, walk forwards covering a marked out 3 meter distance, turn 360° around the 3 meter mark, walk back towards the chair and return to the seated position.
Change in blood pressure (postural hypotension) | Blood pressure will be recorded seven times across three sessions (one week apart) over a period of six weeks throughout the study period.
  Blood pressure will be measured using a fully digitalised blood pressure monitor in sitting and standing. The participants will be asked to remain relaxed with both feet flat on the floor. The blood pressure cuff will be applied around their right bicep, 2.5cm above the elbow joint. The digital screen will then display the systolic and diastolic blood pressure measurements for recording. Blood pressure measurements will be taken before the sitting bout, and after 1 hour, 2 hours and 4 hours.
Change in balance (postural sway) | Postural sway as a measure of static balance will be assessed seven times across three sessions (one week apart) over a period of six weeks throughout the study.
  Postural sway will be assessed using a laser range finder with a 30cm range. The range finder will be attached to the participant when they rise from a chair after the sitting bouts to measure sway.
Change in salivary cortisol | Salivary samples will be collected nine times across three sessions (one week apart) over a period of six weeks to measure cortisol levels in participants.
  This is will be measured by providing a wad of cotton for participants to put in their mouth.
Change in serum inflammatory markers (Venepuncture) | Serum inflammatory markers will be measured six times per participant across three sessions (one week apart) over a period of six weeks throughout the study.
  Blood samples will be collected twice from participants on each of the three visits to measure inflammatory markers.
Change in perception of musculoskeletal comfort | This will be assessed six times for each participant on three sessions (one week apart) over a period of six weeks throughout the study.
  Participants will be asked to rate their level of pain following standing upright, specifically within their lower limb joints, on a scale of 0 (no pain) to 10 (agonising pain).
Change in subjective vitality scale | Vitality will be assessed six times on three occasions (one week apart) over a six-week period throughout the study.
  The Subjective Vitality Scale assesses psychological wellbeing in terms of the subjective feelings of being alive and full of energy, referred to as vitality (Ryan and Frederick, 1997).
Change in Profile of Mood States (POMS) | Participants' mood will be assessed six times on three occasions (one week apart) over a six-week period throughout the study.The questionnaires will be administered before and after each of the three sitting sessions which will be about one week apart.
  The Brief Profile of Mood States (POMS) is a modified shorter version of the Profile of Mood States (McNair, Lorr & Droppleman, 1989). This will be used in the present study as a measure of affective mood. Participants will be instructed to complete the task by rating the 30 mood states, on a scale of 1 (not at all) to 5 (extremely) based on their current mood.
Change in simple reaction time (Simon Task) | This test will be administered six times over a period of six weeks throughout the study. The test will be taken before and after each of the three sitting sessions which will be about one week apart.
  This computer based test assesses cognitive function by creating stimulus- response conflict and measures the participant's capability to respond to the correct stimuli.
Change in Digit Symbol Test score | This test will be taken six times over a period of six weeks throughout the study. The test will be taken twice (before and after 1 hour, 2 hours and 4 hours sitting sessions). The sessions will be about one-week apart.
  This is a computer based measure of cognitive function. The test involves rows containing the symbols in a random order, with empty boxes displayed underneath the symbol. Using the digit-symbol look up table, the participant's task will be to complete the empty digit boxes to match the corresponding symbols, one at a time using the laptop keyboard.
Change in Trial Making Test B score | Trial Making Test B will be administered six times over a period of six weeks throughout the study. The test will be administered before and after each of the three sitting sessions (1 hour, 2 hours and 4 hours). The sessions will be one week apart.
  This cognitive test assesses executive function. It will be completed as a paper version of the Trail Making Test B. The participants will be instructed to complete the test by connecting the numbers and letters in an alternating numerical and alphabetical sequence, by drawing lines between the figures and alphabets (i.e. A, 1, B, 2, etc.) without removing the pen from the paper. Performance will be measured by the time taken to complete the test correctly, therefore the participants will be advised to complete the test as rapidly as possible.
Change in Alice Heim 1&2 test (AH1,2) | AH1,2 will be administered six times over a six week period. The test will be taken before and after each of the three sitting sessions (1 hour, 2 hours and 4 hours). The sessions will be one week apart.
  Alice Heim 1 is the verbal reasoning part of the Alice Heim Group Ability Test (AH4). The section will be preceded by a short practice test . In the Alice Heim 2 test, participants will be instructed to select the most appropriate image based on the instructions given.This is the non-verbal reasoning part of the Alice Heim Group Ability Test (AH4).

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A Greig, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom